CLINICAL TRIAL: NCT04969588
Title: Development and Validation of Kinect Equations to Estimate Body Indices and Body Composition
Brief Title: Kinect Equations for Body Indices and Body Composition
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Principal Investigator, Li-Wen Lee, Consultant Radiologist, Chang Gung Memorial Hospital
Other Study IDs: 202002212A3
Record Dates: First submitted 2021-07-11; First posted 2021-07-20 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Anthropometry; Body Composition
Keywords: Anthropometry; Body Composition
MeSH Terms: interventions — Absorptiometry, Photon

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children and adult: Participants aged 6-65 years old are recruited for the measurements of depth camera, bioelectrical impedance analysis and dual energy X-ray absorptiometry.
  Interventions: Diagnostic Test: Microsoft Azure Kinect Developer Kit; Diagnostic Test: Bioelectrical impedance analyzer; Diagnostic Test: Dual Energy X-ray Absorptiometry

INTERVENTIONS:
Diagnostic Test: Microsoft Azure Kinect Developer Kit — 3D images and 3D joint coordinates are obtained.
Diagnostic Test: Bioelectrical impedance analyzer — Fat mass, fat-free mass and percentage body fat in total body and body segments are estimated.
Diagnostic Test: Dual Energy X-ray Absorptiometry — Skeletal length and body composition are estimated.

SUMMARY:
This perspective observational study will recruited 240 participants for investigating the feasibility of using Microsoft Azure Kinect developer kit as a method for body indices and body composition. Reference methods will be dual energy X-ray absorptiometry and bioelectrical impedance analysis.

DETAILED DESCRIPTION:
The purpose of this research is to validate the precision and accuracy of Microsoft Azure Kinect Developer Kit in the application of body anthropometric index and body composition measures. This study assumes that depth camera along with skeletal tracking package can estimate the 3D joint position and skeletal length. A dual energy X-ray absorptiometry scanner, a medical device with a daily background dose of radiation will be used as the gold standard.

This study aims to investigate the correlation and agreement of using Kinect in estimating skeletal length and body composition in human.A total of 240 participants including children and adults will be recruited for measurements in a 3-year period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children and adult
* Age 6-65 years

Exclusion Criteria:

* Chronic illness or chronic medication use (> 3 months)
* Pregnant
* Metal implant(s) or splint(s)
* Pacemaker implantation
* Limb defect(s) or injury

Ages: 6 Years to 65 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Apparently healthy participants aged 6-65 years are recruited for this study within 3 years. Estimated enrolled number are 240. Eligible participants will visit study site once and take the measurements.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Assess association and agreement in body indices and body composition between Kinect and standard methods. | 36 months
  Correlation and agreement between depth camera results are compared to the results of dual energy X-ray absorptiometry and bioelectrical impedance analysis.
Develop and validate Kinect equations to predict body indices and body composition. | 36 months
  Prediction equations for body indices and body composition are created using dual energy X-ray absorptiometry and bioelectrical impedance analysis as reference tools.

CONTACTS AND LOCATIONS:
Overall Officials: Li-Wen Lee, MD, PhD, Principal Investigator — Chang Gung Memorial Hospital, Chiayi, Taiwan
Locations (1):
- Chang Gung Memorial Hospital, Chiayi City, Taiwan

IPD SHARING:
Plan to Share IPD: No